CLINICAL TRIAL: NCT00182195
Title: A Randomized Trial of a Lung-Open Ventilation Strategy in Acute Lung Injury
Brief Title: Lung Open Ventilation to Decrease Mortality in the Acute Respiratory Distress Syndrome
Acronym: LOVS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hamilton Health Sciences Corporation (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Organization: McMaster University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 38141-1
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2007-04-23 (Estimated); Status verified 2007-04

CONDITIONS: Acute Respiratory Distress Syndrome
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Control Ventilation Strategy

SUMMARY:
A multinational, randomized trial comparing two lung protecting strategies of respiratory life support among critically ill patients with severe lung injury.

DETAILED DESCRIPTION:
To compare an innovative Lung Open Ventilation strategy with a proven low tidal volume strategy, hypothesizing that the Lung Open Ventilation strategy may reduce mortality, other organ dysfunction, and the duration of mechanical ventilation, intensive care, and hospital stay.

ELIGIBILITY:
Inclusion Criteria:

* Invasive mechanical ventilation
* Acute respiratory insufficiency (within past 28 days)
* Bilateral infiltrates on frontal chest radiograph
* Hypoxemia, defined as PaO2/FiO2<=250

Exclusion Criteria:

* Primary cause of respiratory failure is cardiac
* Anticipated duration of mechanical ventilation < 48 hours
* Inability to wean other experimental ventilation strategies
* Severe chronic respiratory disease
* Neuromuscular disease that will prolong mechanical ventilation
* Conditions where hypercapnia-induced intracranial hypertension should be avoided
* Morbid obesity (> 1Kg per cm body weight)
* Pregnancy
* Very unlikely to survive and lack of commitment to life support Underlying irreversible condition with 6 month mortality >= 50%
* Greater than 48 hours elapsed since first eligible
* Current participation in competing trial
* Lack of physician, patient or proxy consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 980
Dates: Start 2000-08; Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Hospital Mortality

SECONDARY OUTCOMES:
Mortality attributed to respiratory failure
Duration of respiratory failure and duration of mechanical failure
Evaluation of respiratory function during mechanical ventilation
Incidence of barotraumas
Non-respiratory organ dysfunction

CONTACTS AND LOCATIONS:
Overall Officials: Maureen O Meade, MD, FRCPC, Principal Investigator — McMaster University
Locations (1):
- Hamilton Health Sciences - General Hospital, Hamilton, Ontario, Canada

REFERENCES:
- [Derived] Mehta S, Cook DJ, Skrobik Y, Muscedere J, Martin CM, Stewart TE, Burry LD, Zhou Q, Meade M. A ventilator strategy combining low tidal volume ventilation, recruitment maneuvers, and high positive end-expiratory pressure does not increase sedative, opioid, or neuromuscular blocker use in adults with acute respiratory distress syndrome and may improve patient comfort. Ann Intensive Care. 2014 Nov 6;4:33. doi: 10.1186/s13613-014-0033-9. eCollection 2014. PMID 25593749
- [Derived] Meade MO, Cook DJ, Guyatt GH, Slutsky AS, Arabi YM, Cooper DJ, Davies AR, Hand LE, Zhou Q, Thabane L, Austin P, Lapinsky S, Baxter A, Russell J, Skrobik Y, Ronco JJ, Stewart TE; Lung Open Ventilation Study Investigators. Ventilation strategy using low tidal volumes, recruitment maneuvers, and high positive end-expiratory pressure for acute lung injury and acute respiratory distress syndrome: a randomized controlled trial. JAMA. 2008 Feb 13;299(6):637-45. doi: 10.1001/jama.299.6.637. PMID 18270352